CLINICAL TRIAL: NCT07399353
Title: Comparative Study Between Fistula Rerouting Technique and Ligation of Intersphincteric Fistula Tract (LIFT) Technique in Treatment of High Perianal Fistula.
Brief Title: Comparative Study: Fistula Rerouting vs. LIFT for High Perianal Fistula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Sedky Ahmed, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-312-2025
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: High Perianal Fistula
Keywords: Fistula rerouting; LIFT (Ligation of Intersphincteric Fistula Tract); High perianal fistula; Anal fistula surgery; Sphincter-saving surgery; Fecal incontinence; Randomized controlled trial
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistula Rerouting Technique Group (Experimental): Participants in this group will undergo a staged Fistula Rerouting procedure. First Stage: The fistulous tract is cored out using diathermy. Dissection is continued until the point where the tract traverses the external anal sphincter. A circumanal incision is made at the anal verge over this point. The intersphincteric space is entered and dissected until the fistulous tract is palpable. The tract is then dissected off the external sphincter via muscle-splitting and transposed into the intersphincteric space. The original defect in the external sphincter is closed with interrupted absorbable sutures. If the transposed tract is too long, its distal portion is excised. A seton may be placed in the new intersphincteric tract to mark it for the second stage, provided this does not risk injury to the mobilized tract.
  Second Stage: After complete healing of the first-stage wound (typically several weeks later), a fistulotomy is performed on the new, transposed intersphincteric tract
  Interventions: Procedure: Fistula Rerouting Technique
- LIFT Technique Group (Experimental): Participants in this group will undergo the Ligation of Intersphincteric Fistula Tract (LIFT) procedure.
  A curvilinear incision is then made in the intersphincteric groove (the groove between the internal and external anal sphincters) overlying the identified tract.
  Dissection proceeds through the intersphincteric plane until the mature, fibrous fistula tract is encountered. The tract is carefully isolated, then divided. Both the internal (toward the anal canal) and external (toward the skin) ends of the divided tract are securely ligated (tied off) with suture material. The infected cryptoglandular tissue surrounding the tract is debrided and removed.
  The internal wound (near the anal canal) and the external wound (in the intersphincteric groove) are debrided and left open to heal by secondary intention, ensuring adequate drainage.
  Interventions: Procedure: Ligation of Intersphincteric Fistula Tract

INTERVENTIONS:
Procedure: Fistula Rerouting Technique — A two-stage, sphincter-preserving surgical procedure for high perianal fistula. Stage 1: The native fistulous tract is surgically dissected and transposed from its trans-sphincteric course into the intersphincteric plane. The defect in the external sphincter is repaired. Stage 2: After complete healing of the first-stage wound, a fistulotomy is performed on the newly created intersphincteric tract. The goal is to eradicate the fistula while minimizing injury to the anal sphincter complex.
  Arms: Fistula Rerouting Technique Group
Procedure: Ligation of Intersphincteric Fistula Tract — A single-stage, sphincter-preserving surgical procedure for perianal fistula. The fistula tract is accessed via an incision in the intersphincteric groove. The tract is identified, dissected, divided, and both ends are ligated. The infected cryptoglandular tissue is excised. The internal and external wounds are debrided and left open to heal by secondary intention. The goal is to close the fistula tract at its origin while preserving sphincter function.
  Arms: LIFT Technique Group

SUMMARY:
The goal of this clinical trial is to compare two different surgery methods for treating a complex type of anal fistula. This condition is an abnormal tunnel connecting the inside of the anus to the skin nearby. The main questions the study aims to answer are:

Which surgery has a lower chance of the fistula coming back (recurrence)?

Which surgery has a lower chance of causing problems with bowel control (incontinence) after healing?

Researchers will compare two surgery groups:

Group 1: Fistula Rerouting Technique - a two-step surgery that moves the fistula tract to a safer area before opening it.

Group 2: LIFT Technique - a surgery that ties off and closes the fistula tract from between the anal muscles.

Participants will be randomly assigned by a computer to one of these two surgery groups. This helps ensure the comparison between the two surgeries is fair.

Participants in this study will:

* Have tests before surgery, including an MRI scan, to confirm they have the specific type of fistula being studied.
* Undergo one of the two planned surgical procedures.
* Attend follow-up visits after surgery at 1 week, 2 weeks, 1 month, and 3 months.
* Be checked during these visits for wound healing, pain, infection, and bowel control.
* Have another MRI scan if the fistula is suspected to have come back.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, parallel-group surgical trial designed to evaluate and compare the efficacy and functional outcomes of two sphincter-preserving techniques for the management of high perianal fistula: the staged Fistula Rerouting Technique (FRT) and the Ligation of Intersphincteric Fistula Tract (LIFT) procedure.

Background and Rationale:

High perianal fistulas, particularly trans-sphincteric and extrasphincteric types, pose a significant surgical challenge. Traditional fistulotomy carries a high risk of postoperative fecal incontinence due to the division of a substantial portion of the anal sphincter complex. Consequently, sphincter-preserving techniques have been developed. The LIFT procedure, introduced in 2007, achieves closure of the fistula tract via an intersphincteric approach. The FRT, described earlier, employs a staged strategy to physically transpose the fistula tract to a safer intersphincteric plane before its division. While both techniques aim to eradicate the fistula while minimizing injury to the continence mechanism, direct comparative evidence regarding their relative effectiveness, recurrence rates, and impact on postoperative continence is lacking in the literature. This trial aims to fill this evidence gap.

Objectives:

The primary objective is to compare the postoperative recurrence rate of high perianal fistula between the FRT and LIFT groups. The secondary objective is to compare the rate of postoperative fecal incontinence between the two techniques. Additional outcomes include time to wound healing, incidence of surgical site infection, postoperative pain scores, patient-reported quality of life related to incontinence, and time to return to normal activities.

Methodology Overview:

Eligible adult patients (aged 20-65 years) diagnosed with a high perianal fistula at Kasr-Alainy Teaching Hospital will be enrolled. Key exclusion criteria include preoperative incontinence, inflammatory bowel disease, and complex branching fistulas. After providing informed consent, participants will undergo preoperative assessment including clinical examination, MRI fistulogram for tract mapping, and baseline continence scoring using the Cleveland Clinic Fecal Incontinence Score (CCFIS).

Participants will be randomly allocated in a 1:1 ratio to either the FRT group or the LIFT group using a computer-generated randomization sequence with allocation concealment.

FRT Group: Participants will undergo the two-stage procedure as described. The second-stage fistulotomy will be performed only after complete healing of the first-stage wound.

LIFT Group: Participants will undergo the single-stage LIFT procedure.

All surgeries will be performed by experienced colorectal surgeons. A standardized postoperative care and follow-up regimen will be applied to all participants, with scheduled assessments at 1 week, 2 weeks, 1 month, 3 months postoperatively. These assessments will include clinical evaluation for recurrence, wound inspection, CCFIS scoring, patient-reported outcome measures, and documentation of any complications or re-interventions. A follow-up MRI will be performed if clinical recurrence is suspected.

Statistical Considerations:

A sample size of 20 patients per group (40 total) has been calculated based on estimates of recurrence rates for high fistulas. Data will be analyzed on an intention-to-treat basis. The findings of this study are expected to provide Level I evidence to help guide surgical decision-making for this complex condition, balancing the goals of fistula eradication and functional preservation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 20-65 years) presenting with a high perianal fistula, defined as:Trans-sphincteric fistula tract traversing the upper two-thirds of the external anal sphincter, Or Extrasphincteric fistula.
* Patients with recurrent perianal fistula.
* Ability to provide informed consent.

Exclusion Criteria:

* Patients with preoperative fecal incontinence (as assessed by the Cleveland Clinic Fecal Incontinence Score).
* Diagnosis of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Pregnant women.
* Pediatric patients (age < 20 years).
* Patients with complex, branching fistula tracts.
* Any contraindication to spinal/general anesthesia or surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fistula Recurrence Rate | Within 3 months after the final surgical procedure
  The proportion of patients in each group with clinically confirmed recurrence of the perianal fistula within 6 months postoperatively. Recurrence is defined as the reappearance of symptoms (pain, discharge) and/or a confirmed tract on postoperative MRI fistulogram.
Postoperative Fecal Incontinence | At 3 months postoperatively
  Change in anal continence status assessed using the Cleveland Clinic Fecal Incontinence Score (CCFIS). The score ranges from 0 (perfect continence) to 20 (complete incontinence). A higher score indicates worse function. Incontinence is defined as a CCFIS ≥ 5.

SECONDARY OUTCOMES:
Time to Complete Wound Healing | From the date of surgery until the date of documented complete healing, assessed up to 3 months
  The number of days required for the surgical wound to heal completely, defined as full epithelialization with no discharge
Postoperative Wound Infection Rate | Within 6 weeks postoperatively
  The proportion of patients in each group developing surgical site infection, defined by the presence of purulent discharge, erythema, warmth, or tenderness requiring antibiotic treatment or intervention.
Postoperative Pain | At 1 week and 2 weeks postoperatively
  Patient-reported pain intensity assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Al-Manial Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No